CLINICAL TRIAL: NCT03476369
Title: A Randomized Controlled Trial of Patients Undergoing Percutaneous Coronary Intervention Who Receive Ticagrelor and Fentanyl
Brief Title: Fentanyl and Crushed Ticagrelor in Percutaneous Coronary Intervention
Acronym: FACTPCI
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Researcher stopped study due to slow accrual rate
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1801-05
Record Dates: First submitted 2018-03-12; First posted 2018-03-26 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Percutaneous Coronary Intervention
MeSH Terms: interventions — Fentanyl; Ticagrelor; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fentanyl and Crushed Ticagrelor (Experimental): Premedicated with Fentanyl (at least 25mcg by IV) followed by Ticagrelor 90mg tablet administered crushed (180 mg dose)
  Interventions: Drug: Fentanyl; Drug: Ticagrelor 90Mg Tablet
- Fentanyl and Non-crushed Ticagrelor (Active Comparator): Premedicated with Fentanyl (at least 25mcg by IV) followed by Ticagrelor 90mg tablet administered as a whole tablet (180 mg dose)
  Interventions: Drug: Fentanyl; Drug: Ticagrelor 90Mg Tablet

INTERVENTIONS:
Drug: Fentanyl — Premedicated with Fentanyl (at least 25mcg by IV)
Drug: Ticagrelor 90Mg Tablet — Ticagrelor administered crushed vs non-crushed

SUMMARY:
During a percutaneous coronary intervention (PCI), Fentanyl is commonly used for sedation. Ticagrelor is also routinely used as anti-platelet agent during PCI. However, a recent study has demonstrated the decrease in effectiveness of Ticagrelor when administered along with Fentanyl. Hence this study was designed to further assess the interaction between crushed vs non crushed Ticagrelor and Fentanyl given during PCI procedures.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing clinically indicated elective or non-elective PCI
* Able to swallow oral medications

Exclusion Criteria:

* Contraindications to ticagrelor or fentanyl (or other opiates)
* Pregnancy
* Any use of P2Y12 inhibitors within 14 days
* Known coagulation disorders
* Pre-procedural treatment with an anticoagulant (oral anticoagulant or low molecular weight heparin)
* Platelet count < 100,000/mm3
* Impaired renal function (Estimated glomerular filtration < 45 ml/min/1.73 m2)
* Impaired hepatic function (Based on medical history)
* Prior or planned transcatheter aortic valve replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Guthrie Clinic, Sayre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fentanyl and Crushed Ticagrelor | Fentanyl and Non-crushed Ticagrelor
Started | 20 | 25
Completed | 16 | 22
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fentanyl and Crushed Ticagrelor | Fentanyl and Non-crushed Ticagrelor | Total
Number analyzed (Participants) | 16 | 22 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.19 (9.58) | 68.50 (8.84) | 67.11 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 13 | 16 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 15 | 22 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 22 | 38
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter] | 31.93 (7.47) | 31.68 (5.76) | 31.79 (6.43)
Smoking status = Former/Current Smoker [Count of Participants; unit: Participants] | 13 | 13 | 26
Diabetes [Count of Participants; unit: Participants] | 8 | 9 | 17
Hypertension [Count of Participants; unit: Participants] | 10 | 18 | 28
Hyperlipidemia [Count of Participants; unit: Participants] | 10 | 17 | 27
Coronary Artery Disease [Count of Participants; unit: Participants] | 11 | 14 | 25
Gastroesophageal Reflux Disease (GERD) [Count of Participants; unit: Participants] | 4 | 8 | 12
Obstructive Sleep Apnea (OSA) [Count of Participants; unit: Participants] | 2 | 1 | 3
Positive Imaging Study [Count of Participants; unit: Participants] — Imaging tests check blood flow to the heart. A positive imaging study shows signs of reduced blood flow or blockages that may cause chest pain or heart attacks. Common tests include stress ultrasound, blood flow scans, CT artery scans, and measurements during heart procedures. These tests help doctors decide if treatment is needed.
  Participants | 7 | 12 | 19
Prior Myocardial Infarction (MI) at Admission [Count of Participants; unit: Participants] | 7 | 9 | 16
Renal Insufficiency [Count of Participants; unit: Participants] | 1 | 2 | 3
Non-Elective Procedure [Count of Participants; unit: Participants] — Percutaneous coronary intervention (PCI) is a procedure used to open blocked or narrowed heart arteries using catheters and related devices. A non-elective procedure is a procedure that was not planned in advance and was performed urgently or as an emergency based on the patient's condition. Patients were classified as non-elective if the procedure was performed due to acute symptoms or findings such as ongoing chest pain, heart attack, unstable angina, or other evidence of reduced blood flow to the heart requiring prompt treatment.
  Participants | 7 | 8 | 15
Primary Procedure Angioplasty Stent Coronary [Count of Participants; unit: Participants] | 16 | 21 | 37
Length of Surgery [Median (Inter-Quartile Range); unit: Hours] | 1.46 [1.26 to 1.95] | 1.40 [1.23 to 1.71] | 1.42 [1.23 to 1.76]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Platelet Function Testing (PFT)-Time Curve (AUC0-6) for the First 6 Hours After the Loading Dose of Ticagrelor
Description: The Platelet Function Testing assay will be VerifyNow Platelet Reactivity Assay which is used institutionally. Results are reported in platelet reactive units (PRUs). Based on previous studies, 208 will be used as an estimated cutoff to distinguish therapeutic and subtherapeutic platelet inhibition, with PRUs equal to or less than 208 being considered therapeutic
Time Frame: 6 hours after the loading dose of Ticagrelor
Population: Not all participants had a test completed at every time.
Measure: Median (Inter-Quartile Range); unit: Platelet Reactive Units (PRUs)/hour
Arm/Group | Fentanyl and Crushed Ticagrelor | Fentanyl and Non-crushed Ticagrelor
Number analyzed (Participants) | 9 | 12
Platelet Reactive Units (PRUs)/hour | 796.34 [420.23 to 950.36] | 622.37 [439.28 to 712.04]

2. Secondary Outcome: In-Hospital Stent Thrombosis
Description: Stent thrombosis while in hospital from time of procedure until discharge
Time Frame: From time of procedure until hospital discharge, up to 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fentanyl and Crushed Ticagrelor | Fentanyl and Non-crushed Ticagrelor
Number analyzed (Participants) | 16 | 22
Participants | 0 | 0

3. Secondary Outcome: In-Hospital Thrombolysis in Myocardial Infarction (TIMI) Major and Minor Bleeding
Description: TIMI bleeding is a standardized clinical trial classification used to grade bleeding severity in cardiovascular studies.
  TIMI major bleeding: Any intracranial hemorrhage, or clinically overt bleeding with a ≥5 g/dL decrease in hemoglobin (or ≥15% absolute drop in hematocrit).
  TIMI minor bleeding: Clinically overt bleeding associated with a 3 to <5 g/dL decrease in hemoglobin (or 10 to <15% absolute drop in hematocrit).
  The measure will assess any participant who had at least a 3 g/dL drop in hemoglobin.
Time Frame: From time of procedure until hospital discharge, up to 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fentanyl and Crushed Ticagrelor | Fentanyl and Non-crushed Ticagrelor
Number analyzed (Participants) | 16 | 22
Participants | 0 | 0

4. Secondary Outcome: In-Hospital Recurrent Myocardial Infarction
Description: Myocardial Infarction while in hospital from time of procedure until discharge
Time Frame: From time of procedure until hospital discharge, up to 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fentanyl and Crushed Ticagrelor | Fentanyl and Non-crushed Ticagrelor
Number analyzed (Participants) | 16 | 22
Participants | 0 | 0

5. Secondary Outcome: In-Hospital Stroke
Description: Stroke while in hospital from time of procedure until discharge
Time Frame: From time of procedure until hospital discharge, up to 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fentanyl and Crushed Ticagrelor | Fentanyl and Non-crushed Ticagrelor
Number analyzed (Participants) | 16 | 22
Participants | 0 | 0

6. Secondary Outcome: In-Hospital Death
Description: Death while in hospital from time of procedure until discharge
Time Frame: From time of procedure until hospital discharge, up to 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fentanyl and Crushed Ticagrelor | Fentanyl and Non-crushed Ticagrelor
Number analyzed (Participants) | 16 | 22
Participants | 0 | 0

7. Secondary Outcome: 30-Day Stent Thrombosis
Description: Stent Thrombosis within 30 days from hospital discharge
Time Frame: 30 days after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Fentanyl and Crushed Ticagrelor | Fentanyl and Non-crushed Ticagrelor
Number analyzed (Participants) | 16 | 22
Participants | 1 | 0

8. Secondary Outcome: 30-Day TIMI Major and Minor Bleeding
Description: as for outcome 3
Time Frame: 30 days after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Fentanyl and Crushed Ticagrelor | Fentanyl and Non-crushed Ticagrelor
Number analyzed (Participants) | 16 | 22
Participants | 0 | 0

9. Secondary Outcome: 30-Day Recurrent Myocardial Infarction
Description: Recurrent myocardial infarction within 30 days after hospital discharge.
Time Frame: 30 days after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Fentanyl and Crushed Ticagrelor | Fentanyl and Non-crushed Ticagrelor
Number analyzed (Participants) | 16 | 22
Participants | 1 | 2

10. Secondary Outcome: 30-Day Stroke
Description: Stroke within 30 days after hospital discharge
Time Frame: 30 days after hospital disharge
Measure: Count of Participants; unit: Participants
Arm/Group | Fentanyl and Crushed Ticagrelor | Fentanyl and Non-crushed Ticagrelor
Number analyzed (Participants) | 16 | 22
Participants | 0 | 0

11. Secondary Outcome: 30-Day All-cause Mortality (Death)
Description: Death within 30 days after hospital discharge
Time Frame: 30 days after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Fentanyl and Crushed Ticagrelor | Fentanyl and Non-crushed Ticagrelor
Number analyzed (Participants) | 16 | 22
Participants | 0 | 0

12. Other Pre Specified Outcome: Hospital Length of Stay
Description: Time (Hours) in the hospital from admission for the procedure until discharge
Time Frame: From admission for the procedure until discharge, assessed up to 3 days
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Fentanyl and Crushed Ticagrelor | Fentanyl and Non-crushed Ticagrelor
Number analyzed (Participants) | 16 | 22
Hours | 27.00 [23.00 to 40.00] | 28.50 [22.25 to 48.75]

13. Other Pre Specified Outcome: 30-Day Hospital Readmission
Description: Readmission to the hospital within 30 days of discharge
Time Frame: 30 days after hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Fentanyl and Crushed Ticagrelor | Fentanyl and Non-crushed Ticagrelor
Number analyzed (Participants) | 16 | 22
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 30 days after hospital discharge
Arm/Group | Fentanyl and Crushed Ticagrelor | Fentanyl and Non-crushed Ticagrelor
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/22
Serious Adverse Events (participants affected / at risk) | 2/16 | 2/22
Other Adverse Events (participants affected / at risk) | 0/16 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fentanyl and Crushed Ticagrelor (N=16) | Fentanyl and Non-crushed Ticagrelor (N=22)
Stent Thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
TIMI bleeding (Blood and lymphatic system disorders) | 0 (0) | 0 (0) — TIMI bleeding is standardized classification to grade bleeding severity in cardiovascular studies. The measure will assess any participant who had at least a 3 g/dL drop in hemoglobin.
Myocardial Infarction (Cardiac disorders) | 1 (1) | 2 (2)
Stroke (Nervous system disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT03476369/Prot_000.pdf
  • Statistical Analysis Plan (2025-12-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT03476369/SAP_001.pdf